CLINICAL TRIAL: NCT06395376
Title: Molecular Networks Involved in the Adaptive Stress Response: The Hot Yoga Study
Brief Title: Adaptive Stress Response: The Hot Yoga Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Floyd Chilton, Professor, Department of Nutritional Sciences Director, Precision Nutrition & Wellness Initiative Associate Director,The BIO5 Institute, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB1911122754
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Inflammation; Aging; Depression, Anxiety
Keywords: Yoga; Hyperthermia; Inflammation; Exercise
MeSH Terms: conditions — Inflammation; Depression; Anxiety Disorders; Hyperthermia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot Yoga Intervention (Experimental): Bikram Hot Yoga intervention: Participants perform a minimum of 60-minutes of Hot Yoga (Bikram Sequence), 3x per week in a heated room (40 degrees C) for 6-weeks
  Interventions: Other: Bikram Hot Yoga Intervention
- Hot Yoga Washout (Other): Hot Yoga Washout: Participants complete a 6-week "Washout" period during which the participants performed no Hot Yoga.
  Interventions: Other: Hot Yoga Washout

INTERVENTIONS:
Other: Bikram Hot Yoga Intervention — Active participants engage in a yoga intervention which entails participating in a minimum of 60-minutes of hot yoga (Bikram sequence), 3x per week in a heated room at 40 degrees C. The intervention will be 6-weeks of active intervention when they are participating in yoga, followed by an 6-week "washout" period where they will be asked to not practice yoga. Participants will be asked to give blood at 9 timepoints throughout the 12-week study, including baseline, week one, midpoint, end of Hot Yoga Intervention (Week 6) and after Washout (Week 12)
  Arms: Hot Yoga Intervention
Other: Hot Yoga Washout — The "Washout" period consists of 6-weeks occurring immediately after the Hot Yoga Intervention during which the participants do not perform any hot yoga.
  Arms: Hot Yoga Washout

SUMMARY:
This is a small intervention study which is aimed at characterizing what is known as the adaptive stress response (also know as "hormesis") in women aged 30-45 years. Participants will perform Bikram Yoga in a room heated to 104°F (40°C) which is often referred to as "Hot Yoga".

The hypothesis of this study is that a protective and health-promoting adaptive stress response can be induced in living humans by performing exercise in a hot environment. The primary question is:How does the body physiologically adapt to performing moderately vigorous exercise in a hot environment?

DETAILED DESCRIPTION:
This is a small scale intervention pilot study which is aimed at characterizing "hormesis" or the "adaptive stress response" in a small cadre (n = 28) of women aged 30-45 years performing moderately vigorous physical activity, Bikram Yoga, in a hot environment, simply referred to as "Hot Yoga". The primary question is:How does the body physiologically adapt to performing moderately vigorous exercise in a hot environment?

The hypothesis of this study which underlies the primary question is that a protective and health-promoting adaptive stress response can be induced in living humans through exposure to mild heat stress and moderately vigorous physical exercise while practicing hot yoga. The central premise is that a combination of environmental stressors during each hot yoga session will induce changes in molecular networks and metabolism that will enhance physical/mental health and physiological resilience.

Primary, secondary and tertiary study endpoints:

Characterize the physiological changes brought on by the adaptive stress response using an "omics" approach. Lipidomics and metabolomics will be used to identify changes in small molecule species found in circulating plasma that are associated with the physiological changes the investigators anticipate will occur with the adaptive stress response.

Characterize the adaptive stress response by measuring the changes in the inflammatory response using common inflammation biomarkers: C-reactive protein (CRP), Tumor Necrosis Factor Alpha (TNF-alpha), and Interleukin-6 (IL-6). A complete blood count (CBC) w/Differential assay will also be performed at baseline and after the last Hot Yoga practice to assess any changes in blood components (red blood cells [RBC], white blood cells [WBC], platelets, etc.) that may have occurred in response to the intervention. In addition, the investigators will use buffy coat to assay all WBCs and will perform both typing and counting of WBCs to assess changes relevant to the adaptive stress response. Finally, buffy coat will be used for DNA isolation to genotype for single nucleotide polymorphisms (SNPs) that are related to the adaptive stress response.

Characterize the acute effect that exercising in a hot environment has on emotional stress and well-being using:

Positive and Negative Affect Schedule - Short Form (PANAS-SF) PROMIS - Global Health Scale

Assess long-term effects of the intervention on emotional stress and well-being using a battery of questionnaires that include Warwick-Edinburgh Mental Well-being Scale (WEMWBS) Patient Health Questionnaire (PHQ-9) Generalized Anxiety Disorder (GAD-7) Perceived Stress Scale (PSS)

Importantly, circulating levels of small molecule metabolites will be determined with metabolomic and lipidomic analyses utilizing HPLC-tandem mass spectrometry. Levels of blood inflammatory and stress biomarkers interleukin-6 (IL-6), Tumor Necrosis Factor Alpha (TNF-α), and C-reactive protein (CRP) will be measured utilizing standard enzyme linked immunosorbent assays (ELISA). These assays may be performed in-house or at Sonora Quest Laboratories.

The investigators will implement the use of biostatistics, bioinformatics, and other statistical methods to analyze, interpret, and express the found data and dependent upon the findings, then use the data as the base for grant funding to conduct a full scale clinical trial testing the aforementioned hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-menopausal women between the aged 30 to 45 years (≥30 years and ≤45 years)
2. Not pregnant/not planning to get pregnant during the study duration
3. Have not previously participated in hot yoga in the last 12-months
4. Able to give informed consent and be willing to participate for the entirety of the study
5. Agree not to take interfering medications (stated in 'Exclusion Criteria' section below) during the duration of the study
6. Agree to allow samples to be stored for future use
7. Pass the preliminary health screening
8. Answer no for every question on the Physical Activity Readiness Questionnaire (PAR-Q ) during preliminary screening

Exclusion Criteria:1) Menopausal 2) Answered "Yes" to any question on the Physical Activity Readiness Questionnaire (PAR-Q) 3) Currently lactating 4) Currently pregnant or plan to get pregnant within the duration of the study 5) Has participated in hot yoga within the last 12-months 6) Used tobacco products (smoked, smokeless, electronic) within the last six months 7) Have diabetes, cancer, heart attack or vascular surgery within the past year, be diagnosed with heart disease, high blood pressure, history of stroke, atherosclerosis, asthma, multiple sclerosis or chronic joint disease 8) Have gallbladder disease or had gallbladder removed 9) Have any of the following health conditions:

* fasting Triglycerides greater than 150 milligrams/deciliter
* Blood pressure greater than 130/90
* Body Mass Index equal to or greater than 30 or less than 19
* Fasting glucose greater than 125 milligrams/deciliter.
* Having a pacemaker or a defibrillator 10) Taking any of the following drugs:
* Taking greater than 100 mg aspirin/day
* Taking non-steroidal anti-inflammatory drugs or oral corticosteroids
* Taking monteleukast-type of allergy medications
* Use of statins, niacin or fibrates or other lipid lowering medications

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Prospective participants need to be healthy women aged 30 and 45 years (≥30 years and ≤45 years). Not pregnant or planning to get pregnant, not lactating, not menopausal.
Enrollment: 20 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | Assessed at baseline, Intervention week1, intervention midpoint (3 weeks), end of intervention (Week 6). end of study (Week 12; after washout)
  cytokines and hsCRP
Blood Lipids | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Lipid panel (milligrams per deciliter, mg/dL)
Hemoglobin A1C | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Comprehensive Metabolic Panel (millimole per mole, mmol/mol)
Fasting glucose/insulin | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Comprehensive Metabolic Panel (milligrams per deciliter, mg/dL)
Immune cell phenotypes | Measured at the Start of Intervention (Week1), intervention midpoint (Week 3), end of intervention (Week 6), and end of study (Week 12; after washout)
  Percent Immune phenotypes

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) (Measures Positive and Negative Mood) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  The Positive and Negative Affect Schedule (PANAS) questionnaire used as a self-report measure of mood and is made up of two mood scales, one measuring positive affect and the other measuring negative affect. The questionnaire consists of 20 items and uses a likert scale of "1" to "5" to measure responses of "1" (Very slightly or not at all), "2" (A little), "3" (Moderately), "4" (Quite a bit), and "5" (Extremely)
PROMIS (Patient Reported Outcomes Measurement Information System) - Global Health Scale (Measures well-being) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  PROMIS is a system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. This instrument uses a "reverse" Likert scale of "5" to "1" to measure responses of "5" (Excellent), "4" (Very good), "3" (Good), "2" (Fair), and "1" (Poor) to measure responses to 10 items.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) (Measures well-being) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) measures subjective well-being and assesses aspects of well-being that are "conducive to happiness or eudemonic" and "sensually self-indulgent or hedonistic". This instrument has 14 items and uses a Likert scale of "1" to "5" to measure responses: "1" (None of the time), "2" (Rarely), "3" (Some of the time), "4" (Often), and "5" (All of the time)
Patient Health Questionnaire (PHQ-9) (Measures depression) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  Patient Health Questionnaire (PHQ-9) is a multipurpose instrument that has two questions (the first is split into 9 "subsections") and is used for screening, diagnosing, monitoring and measuring the severity of depression. A scale of "0-3" is assigned to the four boxes. These numbers represent an individual value for each item (depending on which box is checked) that, when summed, provides a "total score" that is representative of a level of depression.
Generalized Anxiety Disorder (GAD-7) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  Generalized Anxiety Disorder (GAD-7) consists of seven items used to measure worry and anxiety symptoms using a "0" to "3" Likert scale to score responses to "how often": "0" (Not at all sure), "1" (Several Days), "2" (Over half the days), "3" (Nearly every day).
Perceived Stress Scale (PSS) | Assessed at Baseline, Midpoint of Intervention (Week 3), End of Intervention (Week 6) and End of Study (Week 12)
  Perceived Stress Scale (PSS) uses ten questions to measure the degree to which situations in one's life are appraised/perceived as stressful. This instrument uses a Likert scale of "0" to "4": "0" (Never), "1" (Almost never), "2" (Sometimes), "3" (Fairly Often), "4" (Very Often).

OTHER OUTCOMES:
Changes in body wieght | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Body weight in kilograms (kg) will be measured at baseline and at the end of the intervention (Week 6) to determine any changes in body weight as result of participating in the intervention.
Changes Body Mass Index (BMI) in kg/m^2 | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Body Mass Index (BMI, kg/m^2) will be calculated using height measured and baseline and body weight measured at baseline and at the end of intervention (Week 6) to determine any changes in BMI as result of participating in the intervention.
Changes in waist-to-hip ratio (WHR) | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Waist circumference (cm) and hip circumference (cm) will be measured at baseline and end of intervention (Week 8). These measurements will be used to calculate waist-to-hip ratio to determine any changes in WHR as result of participating in the intervention. The ratio is without units.
Changes in blood pressure (Systolic/Diastolic, in mmHg) | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Blood pressure (mmHg) will be measured using an automated blood pressure instrument at baseline and at the end of intervention (Week 6) to determine any changes in blood pressure as result of participating in the intervention.
Change in percent body fat (%Fat) | Measured at Baseline, end of intervention (Week 6), and end of study (Week 12; after washout)
  Body fat (%Fat) was measured using an arm-to-arm bioelectrical impedance analyzer and reported as a percent of total fat relative to total body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Floyd Chilton, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- Tucson Yoga Sol, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No